CLINICAL TRIAL: NCT04329156
Title: Evaluation Of Peri-Implant Emergence Profile Conditioned With Two Different Prosthetic Techniques (Randomized Controlled Clinical Trial)
Brief Title: Evaluation Of Peri-Implant Emergence Profile Conditioned With Two Different Prosthetic Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Dental Public Health clinical instructor and study statistician, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: digital flip vs stock healing
Record Dates: First submitted 2020-03-28; First posted 2020-04-01 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Dental Implants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digitally Flip Technique (Experimental)
  Interventions: Other: Digitally Flip Technique
- Stock Healing Abutment (Active Comparator)
  Interventions: Other: Stock Healing Abutment

INTERVENTIONS:
Other: Digitally Flip Technique — A prefabricated shell will be made then after implant placement, the shell will be attached to a plastic abutment using flowable composite to make a customized healing abutment.
  Arms: Digitally Flip Technique
Other: Stock Healing Abutment — After implant placement, a stock healing abutment will be placed onto the implant and screwed on. It will be selected to be 1-2 mm above the gingival margin and slightly smaller in diameter than the intended final restoration.
  Arms: Stock Healing Abutment

SUMMARY:
The aim of this study is to evaluate and compare two prosthetic conditioning techniques to create natural-like peri-implant emergence profile.

DETAILED DESCRIPTION:
Twenty four patients having a non-restorable tooth will be rehabilitated with flapless immediate implant placement after tooth extraction. The emergence profile will be conditioned with either a stock or a customized healing abutment. A definitive screw retained restoration will be inserted 4 months postoperatively. Peri-implant tissues will be evaluated using pink and white esthetic score, radiographs and periodontal parameters at 3,6 and 12 months after implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Presence of non-restorable maxillary anterior or premolar tooth and its healthy contra-lateral.
* The gingival contour of the tooth to be extracted should be in harmony with the healthy contra-lateral tooth.
* Having thick gingival biotype.

Exclusion Criteria:

* Any medical disorder that could interfere with osseointegration or soft tissue healing.
* Active oral infections or periodontal disease.
* Presence of dehiscence or fenestration defects related to the tooth to be extracted.
* Poor oral hygiene.
* Heavy smokers (>10 cigarette / day).

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-25 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Pink esthetic score (PES) | 3 months
  The PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color and texture. Each variable will be assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score.
Pink esthetic score (PES) | 6 months
  The PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color and texture. Each variable will be assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score.
Pink esthetic score (PES) | 12 months
  The PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color and texture. Each variable will be assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score.
White esthetic score (WES) | 6 months
  The WES is based on five variables of the clinical crown: general tooth form; outline and volume, color, surface texture, translucency and characterization. Each variable will be assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score.
White esthetic score (WES) | 12 months
  The WES is based on five variables of the clinical crown: general tooth form; outline and volume, color, surface texture, translucency and characterization. Each variable will be assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score.
Peri-implant Probing Depth (PD) | 3 months
  Peri-implant probing depth refers to the distance from the gingival margin to the bottom of the sulcus depth. The peri-implant sulcus depth will be measured using a graduated plastic autoclavable periodontal probe. In addition to the aforementioned intervals, it will be measured at the day of final restoration placement. The probe will be held parallel to the long axis of the implant and introduced with light force to the peri-implants sulcus.Measurements will be made at 6 sites around each implant; mesio-buccal, mid-buccal, disto-buccal, mesio-palatal, mid-palatal and disto-palatal. Probing depth of 1 mm or less will be recorded as 1 mm, and those exceeding 1 mm, but less than 2 mm, will be recorded as 2 mm, and so on.
Peri-implant Probing Depth (PD) | 6 months
  Peri-implant probing depth refers to the distance from the gingival margin to the bottom of the sulcus depth. The peri-implant sulcus depth will be measured using a graduated plastic autoclavable periodontal probe. In addition to the aforementioned intervals, it will be measured at the day of final restoration placement. The probe will be held parallel to the long axis of the implant and introduced with light force to the peri-implants sulcus.Measurements will be made at 6 sites around each implant; mesio-buccal, mid-buccal, disto-buccal, mesio-palatal, mid-palatal and disto-palatal. Probing depth of 1 mm or less will be recorded as 1 mm, and those exceeding 1 mm, but less than 2 mm, will be recorded as 2 mm, and so on.
Peri-implant Probing Depth (PD) | 12 months
  Peri-implant probing depth refers to the distance from the gingival margin to the bottom of the sulcus depth. The peri-implant sulcus depth will be measured using a graduated plastic autoclavable periodontal probe. In addition to the aforementioned intervals, it will be measured at the day of final restoration placement. The probe will be held parallel to the long axis of the implant and introduced with light force to the peri-implants sulcus.Measurements will be made at 6 sites around each implant; mesio-buccal, mid-buccal, disto-buccal, mesio-palatal, mid-palatal and disto-palatal. Probing depth of 1 mm or less will be recorded as 1 mm, and those exceeding 1 mm, but less than 2 mm, will be recorded as 2 mm, and so on.
Modified Sulcus Bleeding Index (BI) | 3 months
  A score of 0-3 will be assigned to each labial and palatal surface of the implant then the average for each implant will be calculated according to the following criteria:
  Score 0: No bleeding when a periodontal probe is passed along the gingival margin adjacent to the implant. Score 1: Isolated bleeding spots visible. Score 2: Blood forms a confluent red line on margin. Score 3: Heavy or profuse bleeding.
Modified Sulcus Bleeding Index (BI) | 6 months
  A score of 0-3 will be assigned to each labial and palatal surface of the implant then the average for each implant will be calculated according to the following criteria:
  Score 0: No bleeding when a periodontal probe is passed along the gingival margin adjacent to the implant. Score 1: Isolated bleeding spots visible. Score 2: Blood forms a confluent red line on margin. Score 3: Heavy or profuse bleeding.
Modified Sulcus Bleeding Index (BI) | 12 months
  A score of 0-3 will be assigned to each labial and palatal surface of the implant then the average for each implant will be calculated according to the following criteria:
  Score 0: No bleeding when a periodontal probe is passed along the gingival margin adjacent to the implant. Score 1: Isolated bleeding spots visible. Score 2: Blood forms a confluent red line on margin. Score 3: Heavy or profuse bleeding.
Modified Plaque Index (PI) | 3 months
  The presence or absence of plaque around abutments will be scored at four sites of each implant; buccal, lingual, mesial and distal then the mean will be calculated. This will be carried-out by visual inspection with the aid of a mouth mirror and a plastic periodontal probe after air drying of the abutments. The criteria for assessment include:
  Score 0: No plaque in the gingival area, tested by running the side of plastic probe along the abutment surface at the entrance to the peri-implant sulcus.
  Score 1: Presence of a film of plaque near the gingival margin recognized by running the plastic periodontal probe along the abutment surface.
  Score 2: Moderate accumulation of plaque near or within the peri-implant sulcus, which could be seen naked eye.
  Score 3: Abundant plaque or soft matter within the peri-implant sulcus and or the mucosal sulcus margin and adjacent implant surface.
Modified Plaque Index (PI) | 6 months
  The presence or absence of plaque around abutments will be scored at four sites of each implant; buccal, lingual, mesial and distal then the mean will be calculated. This will be carried-out by visual inspection with the aid of a mouth mirror and a plastic periodontal probe after air drying of the abutments. The criteria for assessment include:
  Score 0: No plaque in the gingival area, tested by running the side of plastic probe along the abutment surface at the entrance to the peri-implant sulcus.
  Score 1: Presence of a film of plaque near the gingival margin recognized by running the plastic periodontal probe along the abutment surface.
  Score 2: Moderate accumulation of plaque near or within the peri-implant sulcus, which could be seen naked eye.
  Score 3: Abundant plaque or soft matter within the peri-implant sulcus and or the mucosal sulcus margin and adjacent implant surface.
Modified Plaque Index (PI) | 12 months
  The presence or absence of plaque around abutments will be scored at four sites of each implant; buccal, lingual, mesial and distal then the mean will be calculated. This will be carried-out by visual inspection with the aid of a mouth mirror and a plastic periodontal probe after air drying of the abutments. The criteria for assessment include:
  Score 0: No plaque in the gingival area, tested by running the side of plastic probe along the abutment surface at the entrance to the peri-implant sulcus.
  Score 1: Presence of a film of plaque near the gingival margin recognized by running the plastic periodontal probe along the abutment surface.
  Score 2: Moderate accumulation of plaque near or within the peri-implant sulcus, which could be seen naked eye.
  Score 3: Abundant plaque or soft matter within the peri-implant sulcus and or the mucosal sulcus margin and adjacent implant surface.
Radiographic evaluation of alveolar bone using cone beat computed tomography (CBCT) | 3 months
  The level of alveolar bone around each implant will be assessed using CBCT. The vertical bone change (distance from the implant platform to the first bone-to-implant contact, in mm) around each implant will be assessed at the buccal, lingual, mesial and distal aspects then the mean will be calculated.
Radiographic evaluation of alveolar bone using cone beat computed tomography (CBCT) | 6 months
  The level of alveolar bone around each implant will be assessed using CBCT. The vertical bone change (distance from the implant platform to the first bone-to-implant contact, in mm) around each implant will be assessed at the buccal, lingual, mesial and distal aspects then the mean will be calculated.
Radiographic evaluation of alveolar bone using cone beat computed tomography (CBCT) | 12 months
  The level of alveolar bone around each implant will be assessed using CBCT. The vertical bone change (distance from the implant platform to the first bone-to-implant contact, in mm) around each implant will be assessed at the buccal, lingual, mesial and distal aspects then the mean will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Badee, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Mohamed M Khamis, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Ahmed A Abdelhakim, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Rania Abdelaziz, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt